CLINICAL TRIAL: NCT00992121
Title: An Open-Label Study to Investigate the Pharmacodynamics of a Repeat Dose Regimen of Bevacizumab (10 mg/kg q2w) and Escalating Repeat Doses of Pazopanib in Renal Cell Carcinoma
Brief Title: An Open-Label Pharmacodynamic Study of Bevacivumab and Pazopanib in Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 111687
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Carcinoma, Renal Cell
Keywords: pazopanib; Renal Cell Carcinoma; Kidney; cancer; bevacizumab
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms | interventions — Bevacizumab; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part I and 2 week dosing Part II (Other): Part I - bevacizumab 3 infusions at 2 week intervals Part II - pazopanib dosing 2 weeks in 3-week cycles
  Interventions: Drug: Bevacizumab; Drug: Pazopanib 2 week
- Part I and 3 week dosing Part II (Other): Part I - bevacizumab 3 infusions at 2 week interval, Part II - pazopanib dosing 3 weeks in 3-week cycles
  Interventions: Drug: Bevacizumab; Drug: Pazopanib 3 week

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab - 3 infusions of 10mg/kg administered at 2 week intervals - Part I
Drug: Pazopanib 2 week — Pazopanib for first 2 weeks of each 3-week cycles as follows: 1) 200 mg twice weekly, 2) 200 mg every other day, 3) 200 mg qd, 4) 400 mg qd, 5) 800 mg qd, and 6) 1200 mg qd (Group 1).
  Maintenance pazopanib 800 mg qd for all 3 weeks throughout repeating 3-week cycles. Number of cycles: until death, loss of clinical benefit, unacceptable toxicity, or withdrawal from the study for other reasons.
  Arms: Part I and 2 week dosing Part II
Drug: Pazopanib 3 week — Pazopanib throughout each 3-week cycle as follows: 1) 200 mg twice weekly, 2) 200 mg every other day, 3) 200 mg qd, 4) 400 mg qd, 5) 800 mg qd, and 6) 1200 mg qd (Group 1).
  Maintenance pazopanib 800 mg qd for all 3 weeks throughout repeating 3-week cycles. Number of cycles: until death, loss of clinical benefit, unacceptable toxicity, or withdrawal from the study for other reasons.
  Arms: Part I and 3 week dosing Part II

SUMMARY:
This study will determine whether blood tests, tumour imaging and tumour tissue analysis can reveal effects of drugs that block blood vessel growth (angiogenesis) in patients with renal cancer.

DETAILED DESCRIPTION:
This single-centre, two-part, open-label study is designed to evaluate pharmacodynamic (PD) effects of bevacizumab and pazopanib in subjects with renal cancer who experience disease progression following at least one prior therapy of documented clinical benefit. In Part I, subjects will receive 3 infusions of 10 mg/kg bevacizumab, administered at 2-week intervals. The PD response to bevacizumab will be evaluated over 6 weeks using imaging techniques (magnetic resonance imaging; computed tomography [CT]; and positron emission tomography), intratumoural VEGF signaling by immunohistochemisty, plasma and serum biomarkers, and circulating tumour cells. Subjects may continue into Part II if, in the opinion of the investigator, the subject would derive continued clinical benefit from anti-angiogenic therapy. In Part II, each subject will receive sequentially escalating doses of oral pazopanib in 3-week cycles as follows: 1) 200 mg twice weekly, 2) 200 mg every other day, 3) 200 mg daily, 4) 400 mg daily, 5) 800 mg daily, and 6) 1200 mg daily. Subjects entering Part II will be randomised to receive treatment either throughout each 3-week cycle (Group 1) or for the first 2 weeks of each cycle only, followed by a 1 week treatment holiday (Group 2). After completion of Part II dose escalation subjects will receive continuous pazopanib at a dose of 800 mg daily in repeating 3-week cycles. These subjects will receive pazopanib until loss of clinical benefit, death, unacceptable toxicity, or withdrawal from the study for other reasons.

ELIGIBILITY:
Inclusion Criteria:

* Histologically (any histological subtype) or cytologically confirmed unresectable RCC with a clear cell component.
* Experienced documented evidence of radiological progression based on Response Evaluation Criteria in Solid Tumors [RECIST] while on first line (or greater) RCC therapy and within 6 months prior to the first dose of study medication (bevacizumab).
* Evidence of unidimensionally measurable disease (i.e., at least 1 malignant tumour mass that can be accurately measured in at least 1 dimension with the longest diameter greater than or equal to 20 mm with conventional CT or MRI or V10 mm with spiral CT scan [if spiral CT scan is used, minimum lesion size should be twice the reconstruction interval used, e.g., if reconstruction size is 7 mm, lesion size should be greater than or equal to 14 mm]) Note: Subject should be excluded if all baseline measurable lesions are within previously irradiated areas.
* Free of any malignant disease other than RCC for at least 5 years prior to the first dose of study medication (bevacizumab) in this study, with the exception of the following: Cervical carcinoma in situ, Melanoma in situ, Basal or squamous cell carcinoma of the skin
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1
* Resolution of all acute toxic effects of prior chemotherapy, radiotherapy, or surgical procedures to NCI CTCAE Grade 1 or less.
* Adequate organ function as defined by laboratory ranges Note: Laboratory values just outside of these ranges may be included if in the view of the investigator and medical monitor, these findings will not interfere with the study or pose an unacceptable risk to the subject.
* Capable of giving written informed consent, and willing and able to comply with the requirements and restrictions listed in the consent form.
* Males and females greater than or equal to 18 years of age at screening. A female subject is eligible to participate if she is of non-childbearing potential (see below) or if she is of childbearing potential and agrees to use one of the defined contraception methods from the time of first dose of study medication (bevacizumab) until 4 months after the last dose of study medication (bevacizumab or pazopanib).

Non-childbearing potential is defined as pre-menopausal females with a documented bilateral tubal ligation, bilateral oophorectomy, or hysterectomy; or postmenopausal females with 12 months of spontaneous amenorrhea. If the exact duration of amenorrhea is unknown, a blood sample with simultaneous follicle stimulating hormone (FSH) greater than or equal to 40 MIU/mL and estradiol less than or equal to 40 pg/mL (less than or equal to 140 pmol/L) will be required as confirmation. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the approved contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.

A male subject is eligible to participate if he agrees to use one of the contraception methods listed in from the time of first dose of study medication (bevacizumab) until 4 months after the last dose of study medication (bevacizumab or pazopanib).

Inclusion criteria for progression to Part II

* The subject met all eligibility criteria (inclusive of inclusion and exclusion criteria) for participation in Part I of the study.
* In the opinion of the Investigator, the subject would derive continued therapeutic benefit from anti-angiogenic therapy.
* In the opinion of the Investigator, there are no safety concerns that would present an unacceptable benefit:risk profile for treatment with pazopanib.
* The subject is able to swallow and retain oral medication.

Exclusion Criteria:

* Clinical evidence of cancer metastatic to the central nervous system or leptomeningeal carcinomatosis.
* Previous treatment with bevacizumab or pazopanib, either alone or in combination with other therapy.

Note: Patients who have previously received treatment with cytokine or anti-angiogenic agents other than bevacizumab and pazopanib may be considered for the study.

* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to bevacizumab or pazopanib or components of bevacizumab or pazopanib (other than active drugs), or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates participation.
* Any other anticancer therapy (radiotherapy, chemotherapy, or immunotherapy) within 28 days prior to the first dose of study medication and extending through completion of treatment and all study procedures. Prior palliative radiotherapy to metastatic lesion(s) is permitted, provided there is at least one measurable lesion that has not been irradiated.
* Use of an investigational agent, including an investigational anti-cancer agent, within 28 days or 5 half-lives, whichever is longer, prior to the first dose of study medication.
* Assessable disease is unsuitable for biopsy or the patient is unwilling or not sufficiently fit to undergo serial biopsies of their cancer at the time points specified in Section 4.7.
* A major surgical procedure or traumatic injury within 28 days prior to the first dose of study medication (bevacizumab), or anticipation of a major surgical procedure (that cannot be rescheduled) from the first dose of study mediciation through 28 days after the last dose of study medication. The investigator should confirm that any prior surgical incision has fully healed prior to initiating treatment.
* Evidence of active bleeding or bleeding diathesis, or any serious, non-healing wound, ulcer, or bone fracture.
* Hemoptysis within 6 weeks of the first dose of study medication.
* Use of therapeutic doses of warfarin within 5 half-lives of the first dose of study medication and during treatment in the study. Note: Use of low molecular weight heparin is permitted during the study. Patients may be switched from warfarin to low molecular weight heparin for the duration of this study if, in the opinion of the Investigator, doing so does not present an undue safety risk to the patient.
* National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 hemorrhage within 28 days of the first dose of study medication.
* Clinically significant gastrointestinal abnormalities including, but not limited to: Malabsorption syndrome, Major resection of the stomach or small bowel that could affect the absorption of study drug, Active peptic ulcer disease, Known intraluminal metastatic lesion(s) with suspected bleeding, Inflammatory bowel disease, Ulcerative colitis, or other gastrointestinal conditions with increased risk of perforation, History of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess, or symptomatic diverticulitis within 28 days of the first dose of study medication (bevacizumab).
* Known endobronchial lesions or involvement of large pulmonary vessels by tumor.
* Active or uncontrolled infection at the time of first dose of study medication (bevacizumab) that, in the opinion of investigator, is clinically significant and presents a safety risk to participation in the study.
* Prolongation of corrected QT interval (QTc) >480 milliseconds (msec).
* Previous positive test result for human immunodeficiency virus (HIV) antibody, as determined on medical history.
* Any of the following within 6 months prior to the first dose of study medication (bevacizumab): Cardiac angioplasty or stenting, Severe and/or unstable angina, Myocardial infarction, Coronary artery bypass graft (CABG), Class III or IV congestive heart failure (as defined by the New York Heart Association [NYHA]), Symptomatic peripheral vascular disease, Cardiac dysrhythmias of NCI CTCAE Grade 2 or greater and atrial fibrillation of any grade.
* History of cerebrovascular accident or transient ischemic attack
* Poorly controlled hypertension, defined as systolic blood pressure (SBP) of geater than or equal to 140 mmHg or diastolic blood pressure (DBP) of geater than or equal to 90 mmHg.

Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. If antihypertensive medications are initiated or adjusted, blood pressure must be re-assessed on two occasions that are separated by a minimum of 24 hours. The SBP/DBP values from each blood pressure assessment must be geater than 140/90 mmHg in order for a subject to be eligible for the study.

* History of pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible. As stated above, warfarin should not be administered within 5 half-lives of the first dose of study medication.
* Internal metal medical devices or other metal items that may place the subject's health at risk and/or interfere with MRI scans, including cardiac pacemakers, aortic or cerebral aneurysm clips, artificial heart valves, ferromagnetic implants, shrapnel, wire sutures, joint replacements, bone or joint pins/rods/screws/clips, or non-removable metal jewellery (e.g., rings).
* History of hypersensitivity to gadolinium or other intravenous dye contrast agents.
* History of hypersensitivity to iodine-based contrast agents or history of severe asthma.
* Subjects with type II diabetes who are currently receiving metformin therapy and, in the judgement of the investigator, would be unable to forego therapy for an approximate 24-hour period around each [18F]FDG-PET procedure.
* Any other acute or chronic medical condition or abnormality (e.g., laboratory abnormality) that, in the opinion of the investigator, may result in an unacceptable safety risk to the subject from participation in this study (either due to bevacizumab, pazopanib, or study procedures) or may interfere with the interpretation of the subject's data, and therefore would make the subject inappropriate for entry in this study.
* Pregnant females, as determined by positive serum Beta-hCG test at screening.
* Lactating females who are unwilling to discontinue nursing from the time of first dose of study medication (bevacizumab) through 4 months after the last dose of study medication (bevacizumab or pazopanib).
* Any serious and/or unstable pre-existing medical, psychiatric, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-11-18 (Actual); Primary Completion 2013-11-01 (Actual); Study Completion 2013-11-01 (Actual)

PRIMARY OUTCOMES:
Tumour size, as measured by the sum of the longest diameters of all target lesions on CT | 6 weeks

SECONDARY OUTCOMES:
Plasma levels of pharmacodynamic markers of study drug effect | 6 weeks Part I; 15 weeks Part II; 6 weeks during maintenance therapy

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- See also: Results for study 111687 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/111687?search=study&search_terms=111687#rs